CLINICAL TRIAL: NCT00906152
Title: Study of the Association Between Low Back Pain and the Quality of Sleep
Brief Title: Association Between Low Back Pain and Quality of Sleep
Status: Completed | Type: Observational
Sponsor: Kovacs Foundation (Other)
Responsible Party: Principal Investigator, Francisco M. Kovacs, Director of Scientific Department, Kovacs Foundation, Kovacs Foundation
Other Study IDs: FK-29
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2014-03-13 (Estimated); Status verified 2014-03

CONDITIONS: Quality of Sleep; Subacute or Chronic Low Back Pain; Disability; Catastrophizing; Depression
Keywords: quality of sleep; low back pain; disability; catastrophizing; depression
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Low Back Pain

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Subacute low back pain; chronic low back pain: Patients with subacute or chronic low back pain seen in the Primary Care Centers participating in the study.

SUMMARY:
A prospective study to assess the association between the change in quality of sleep and the change in intensity of pain in Spanish patients seen for subacute or chronic low back pain. The objective is to determine the prevalence of sleep alterations, the association between quality of sleep and intensity of pain, degree of disability, intensity of catastrophizing and depression.

ELIGIBILITY:
Inclusion Criteria:

* patients with non-specific low back pain of more than 14 days duration
* seen in health centers participating in the study
* who accept to participate and sign the consent form
* without age limits and regardless of gender

Exclusion Criteria:

* inability to complete the questionnaires (illiteracy, dementia)
* inflammatory rheumatologic disease, fibromyalgia, cancer in last 5 years

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients seen for low back pain in the primary care centers participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 437 (Actual)
Dates: Start 2009-09; Primary Completion 2012-08 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Assessment of the association between low back pain and quality of sleep in patients with subacute or chronic low back pain. | 3 months

SECONDARY OUTCOMES:
Assessment of the association between quality of sleep and disability, catastrophizing and depression in patients with subacute or chronic low back pain. | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Francisco M Kovacs, MD, PhD, Study Director — Kovacs Foundation, Palma de Mallorca, 07012, Spain; Víctor Abraira, PhD, Principal Investigator — Hospital Ramón y Cajal, Unidad de Bioestadística Clínica, Madrid, Spain
Locations (2):
- Spain (2):
  - Kovacs Foundation, Palma de Mallorca, Balearic Islands
  - Hospital Ramón y Cajal, Madrid, Madrid

REFERENCES:
- [Background] Hansson EK, Hansson TH. The costs for persons sick-listed more than one month because of low back or neck problems. A two-year prospective study of Swedish patients. Eur Spine J. 2005 May;14(4):337-45. doi: 10.1007/s00586-004-0731-3. Epub 2004 May 19. PMID 15150703
- [Background] Moldofsky H. Sleep and pain. Sleep Med Rev. 2001 Oct;5(5):385-396. doi: 10.1053/smrv.2001.0179. PMID 12531004
- [Background] Tang NK, Wright KJ, Salkovskis PM. Prevalence and correlates of clinical insomnia co-occurring with chronic back pain. J Sleep Res. 2007 Mar;16(1):85-95. doi: 10.1111/j.1365-2869.2007.00571.x. PMID 17309767